CLINICAL TRIAL: NCT05917301
Title: PROspective Phase II Trial of Pre-operative Hypofractionated protoN Therapy for Extremity and Truncal Soft Tissue sarcOma
Brief Title: Pre-operative Hypofractionated Proton Therapy
Acronym: PRONTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Robert L. Sloan Fund for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIB2289; IRB00335181 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2023-06-01; First posted 2023-06-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: proton therapy; soft tissue sarcoma; hypofractionated
MeSH Terms: conditions — Sarcoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-operative hypofractionated proton therapy (Experimental): Patients will have 5 fractions of proton therapy prior to surgical resection of their sarcoma.
  Interventions: Radiation: hypofractionation

INTERVENTIONS:
Radiation: hypofractionation — This study is being done to see if hypofractionation in treating sarcoma, will also provide patients with a faster and safer treatment outcome.

SUMMARY:
This study is being done to examine whether proton therapy for certain kinds of sarcomas (extremity and trunk soft tissue) is safe and effective. As part of the study, patients will have five fractions of proton therapy before the participants have surgery for the sarcoma. The study will measure wound complications and functional outcomes / quality of life after the procedures.

Patients will be asked to complete questionnaires about the treatment and quality of life from the time of enrollment until about two years after surgery. Otherwise, the participants will have standard of care follow ups with the treatment team.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* Patients with primary or locally recurrent extremity or truncal soft tissue sarcoma
* WHO/ECOG status ≤2

Exclusion Criteria:

* History of prior local radiation therapy
* Inability to tolerate treatment position for duration of simulation or treatment
* Tumor originating in retroperitoneal location
* Patients planned for systemic therapy including chemotherapy, targeted agents, and immunotherapy
* Co-existing malignancy or treated malignancy in the last 2 years expected to limit life expectancy; does not include completely resected cutaneous basal cell carcinoma, squamous cell carcinoma, in situ breast or cervical malignancies, or other pathologies at the discretion of the investigators.
* Confirmed pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Rate of major wound complications | 90 days after surgery
  Number of major wound complications as defined by the CAN-NCIC-SR2 trial ("secondary operation under general or regional anaesthesia for wound repair (debridement, operative drainage, and secondary wound closure including rotationplasty, free flaps, or skin grafts), or wound management without secondary operation…[including] an invasive procedure without general or regional anaesthesia (mainly aspiration of seroma), readmission for wound care such as intravenous antibiotics, or persistent deep packing for 120 days or longer.")

SECONDARY OUTCOMES:
Incidence of acute grade ≥3 adverse events | 2 years after treatment
  Rate of acute grade 3 or higher adverse events (CTCAE5)
Rate of local recurrence free survival | 1 and 2 years after enrollment
  Number of patients without local recurrence on CT and/or MRI at specified time points.
Rate of metastasis free survival | 1 and 2 years after enrollment
  Number of patients without metastasis on CT and/or MRI at specified time points.
Rate of late grade ≥2 radiation toxicity | median two year follow up
  Rate of grade 2 or higher CTCAE5 adverse events associated with radiation therapy (fibrosis, lymphedema, or joint stiffness).
Musculoskeletal Tumor Rating Scale scores | baseline, 2-12 weeks after end of radiation therapy, after surgery (3-6 month follow up), every 3 months during follow up for 2 years
  The Musculoskeletal Tumor Rating Scale measures physical function in patients with musculoskeletal tumors. The total score for the MSTS ranges 0-30 with higher scores indicating better function.
Toronto Extremity Salvage Score (TESS) scores | baseline, 2-12 weeks after end of radiation therapy, after surgery (3-6 month follow up), every 3 months during follow up for 2 years
  The Toronto Extremity Salvage Score (TESS) measures physical function in patients with musculoskeletal tumors. The total score for the TESS ranges 0-100 with higher scores indicating better function.
Functional Assessment of Cancer Therapy-General (FACT-G) scores | baseline, 2-12 weeks after end of radiation therapy, after surgery (3-6 month follow up), every 3 months during follow up for 2 years
  The Functional Assessment of Cancer Therapy-General (FACT-G) measures quality of life for patients with cancer. The total score for the FACT-G ranges 0-108 with higher scores indicating better function.
Rate of pathologic complete response | through study conclusion (estimated 5 years from opening)
  Pathologic complete response rate is reported as the number of patients who achieve pathologic complete response after treatment.
  As per the NCCN guidelines, pathologic response is graded by the system recommended by the AJCC Cancer Staging Manual and CAP guidelines:
  Complete response - no remaining viable cancer cells Moderate response - only small clusters/single cancer cells remain Minimal response - residual cancer remaining, but with predominant fibrosis Poor response - minimal/no tumor kills, extensive residual cancer

CONTACTS AND LOCATIONS:
Overall Officials: Curtland Deville, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Gogineni E, Chen H, Hu C, Boudadi K, Engle J, Levine A, Deville C Jr. Prospective phase II trial of preoperative hypofractionated proton therapy for extremity and truncal soft tissue sarcoma: the PRONTO study rationale and design. Radiat Oncol. 2024 May 14;19(1):56. doi: 10.1186/s13014-024-02447-0. PMID 38745333